CLINICAL TRIAL: NCT07169513
Title: Targeting the Inflammasome With Anti-platelet Therapy: A Mechanistic Study
Brief Title: Mechanistic Study of Anti-Platelet Therapy in Atherosclerosis
Acronym: MPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 174661
Record Dates: First submitted 2025-07-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Arterial Disease; Silent Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: The study is a randomised, single-blind, controlled crossover trial in two groups of patients following treatment with aspirin and clopidogrel; (1) patients with abnormally high carotid intima-media thickness (cIMT) - defined by an intima-media thickness (IMT) above the 75th centile for age and sex; and (2) patients with a confirmed diagnosis of PAD (ankle-brachial index below 0.9) with Rutherford classification grade of 1-3.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin/Clopidogrel (Active Comparator)
  Interventions: Drug: Aspirin 75 mg daily; Drug: Clopidogrel 75 mg daily
- Clopidogrel/DAPT (Active Comparator)
  Interventions: Drug: Clopidgrel 75 mg daily; Drug: Aspirin 75 mg daily + Clopidgrel 75 mg daily

INTERVENTIONS:
Drug: Aspirin 75 mg daily — For group 1 patients
  Arms: Aspirin/Clopidogrel
Drug: Clopidogrel 75 mg daily — For group 2 patients
  Arms: Aspirin/Clopidogrel
Drug: Clopidgrel 75 mg daily — For group 1 patients
  Arms: Clopidogrel/DAPT
Drug: Aspirin 75 mg daily + Clopidgrel 75 mg daily — For group 2 patients
  Arms: Clopidogrel/DAPT

SUMMARY:
Many people have a higher chance of getting heart problems. These individuals include people who are very overweight (obesity), have high blood pressure (hypertension), diabetes, or other health concerns. Heart problems often happen because of a condition called atherosclerosis. This condition is when the arteries, which are the blood vessels carrying blood from the heart, become hard and inflamed (swollen and irritated) at the same time. Atherosclerosis causes arteries narrowing, making it harder for blood to flow through. The signs of atherosclerosis can be mild, like feeling chest pain (called angina) because the heart isn't getting enough blood. In more serious cases, it can lead to a heart attack.

Think of inflammation as the body's natural alarm system. When a person gets hurt or sick, the body releases special chemicals. These chemicals tell the immune system (the body's defence team) to come and help. Their job is to heal the injury or fight off the infection.

While inflammation is usually good, sometimes it can go wrong. Atherosclerosis is one of these conditions where the inflammation in the blood vessels becomes abnormal. This ongoing inflammation can harm the body and lead to various heart problems and other health issues not directly related to the heart.

In atherosclerosis, platelets (cell fragments in our blood that form clots and stop or prevent bleeding) bind to monocytes (a type of white blood cell and a type of phagocyte - part of the immune system) to form clusters called monocyte platelet aggregate (MPA). Studies have shown that people with atherosclerosis have higher levels of the monocytes clustering with the platelets. This aggregate contributes to the worsening of atherosclerosis. Additionally, this aggregate can predict the risk of developing various cardiac diseases.

Anti-platelet (anti-clotting) medications work by stopping platelet function. In this study, investigators are giving participants two different anti-platelet medications to study the effect of these medications on the level of MPA. The target people of our study are the people with silent atherosclerosis (there is an accumulation of lipids in the blood vessels but no signs or symptoms). No existing research demonstrates whether the two most commonly prescribed anti-platelets (aspirin and clopidogrel) can help reduce MPA levels. This study aims to show the effect of anti-platelet medications on the level of MPA and other inflammatory indicators. The two medications are aspirin and clopidogrel. These two drugs are already available in the market and widely used by different patients for different reasons. Aspirin and clopidogrel have different modes of action to stop platelet function.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Male or female age 18 years or older
* Willing to participate in the study, and able to give informed consent
* Negative pregnancy test for a childbearing age woman
* Receiving standard of care
* Confirmed atherosclerotic cardiovascular risk based on clinical assessment

Group 2:

* Male or female age 18 years or older
* Willing to participate in the study, and able to give informed consent
* Receiving standard of care
* Negative pregnancy test for a childbearing age woman
* Confirmed diagnosis of peripheral arterial disease (ankle-brachial index below 0.9) with Rutherford grade 1-3.

Exclusion Criteria:

Group 1:

* Diabetes
* Receiving any anti-platelet medications within the last two weeks
* Receiving any anticoagulant medications within the last two weeks
* Receiving statin medications within the last two weeks
* Known major organ dysfunction
* Significant co-morbidities
* Pregnancy or lactating woman
* Unwilling, or unable to give informed consent
* Presence of co-existing autoimmune disease
* Hypersensitivity to aspirin or clopidogrel
* Severe hepatic impairment (Child-Pugh grade C)
* Active peptic ulcer
* Presence of co-existing inflammatory or autoimmune diseases
* Frequent use of medications known to affect platelet function five days before baseline phlebotomy and during the study

  * Non-steroidal anti-inflammatory drugs (NSAIDs)
  * Antihistamines
  * Selective serotonin reuptake inhibitors
* Platelet count < 100 × 109 /L or > 450 × 109 /L
* Anaemia
* Any known bleeding diathesis
* Currently involved in other clinical research studies

Group 2:

* Diabetes
* Patients with PAD Rutherford category of more than 3
* Receiving any anticoagulant medications within the last two weeks
* Known major organ dysfunction
* Pregnancy or lactating woman
* Unwilling, or unable, to give informed consent
* Hypersensitivity to aspirin or clopidogrel
* Severe hepatic impairment (Child-Pugh grade C)
* Active peptic ulcer
* Presence of co-existing autoimmune disease
* Frequent use of medications known to affect platelet function five days before baseline phlebotomy and during the study

  * Non-steroidal anti-inflammatory drugs (NSAIDs)
  * Antihistamines
  * Selective serotonin reuptake inhibitors
* Platelet count < 100 × 109 /L or > 450 × 109 /L
* Anaemia
* Any known bleeding diathesis
* Currently involved in other clinical research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Monocyte-platelet aggregates (MPAs) | Maximum 14 weeks
  Changes in the percentages of monocyte-platelet aggregates (MPAs) in two groups of patients following treatment with aspirin and clopidogrel using flow cytometry

SECONDARY OUTCOMES:
Monocyte and platelet activation/phenotype | Maximum 14 weeks
  Measure the effect of aspirin, clopidogrel, and their combination on monocyte and platelet activation/phenotype using flow cytometry
Circulating mediators of inflammation | Maximum 14 weeks
  Measure the influence of aspirin, clopidogrel, and their combination on the level of circulating mediators of inflammation using multiplex Luminex assay
Gene expression | Maximum 14 weeks
  Determine how aspirin, clopidogrel, and their combination modulate gene expression using single-cell RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No